CLINICAL TRIAL: NCT05397730
Title: Levels of Mycobacterium Tuberculosis Cell-free DNA (MTB cfDNA) in Tuberculous and Non-tuberculous Pleural Effusion
Brief Title: MTB cfDNA Levels in TBP
Acronym: MYDNITE
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ka Pang Chan, Doctor (Clinical Lecturer), Chinese University of Hong Kong
Other Study IDs: TBP_cfDNA_levels
Record Dates: First submitted 2022-05-23; First posted 2022-05-31 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Tuberculosis, Pleural
Keywords: Tuberculosis, Tuberculous pleuritis, cell-free DNA
MeSH Terms: conditions — Tuberculosis, Pleural; Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Pleural fluid and blood obtained from patients with TBP and non-TBP will be stored for subsequent analysis using genetic sequencing techniques.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TBP: Patients with definite or probable tuberculous pleuritis
  Interventions: Diagnostic Test: Mycobacterium tuberculosis (MTB) cell-free DNA (cf-DNA)
- Non-TBP: Patients without tuberculous pleuritis
  Interventions: Diagnostic Test: Mycobacterium tuberculosis (MTB) cell-free DNA (cf-DNA)

INTERVENTIONS:
Diagnostic Test: Mycobacterium tuberculosis (MTB) cell-free DNA (cf-DNA) — Comparing the diagnostic accuracy between MTB cfDNA and PCR on diagnosing tuberculous pleuritis
  Other Names: Mycobacterium tuberculosis PCR

SUMMARY:
Tuberculous pleuritis (TBP) is the most common manifestation of extrapulmonary TB. Its diagnosis is challenging due to the low sensitivity of mycobacterial culture from the pleural fluid and the need for invasive pleural biopsy. Preliminary data has shown the superior sensitivity of Mycobacterium tuberculosis cell-free DNA (MTB cfDNA) to conventional culture and MTB polymerase chain reaction (PCR), but the cutoff level of MTB cfDNA was not determined. This study involves a prospective collection of pleural fluid due to TBP and non-TBP aetiologies, with subsequent testing by MTB culture, MTB cfDNA and MTB PCR. The levels of MTB cfDNA in the pleural fluid will be correlated with different types of diagnosis, and its diagnostic accuracy will be compared with conventional culture and MTB PCR. A confirmatory study result of MTB cfDNA can shorten the time to diagnosis, reduce the need for pleural biopsy and prevent the delay of definitive treatment.

DETAILED DESCRIPTION:
Tuberculosis (TB) is one of the major global health threats, with an estimated global incidence of 9.87 million cases in 2020 and it is the second leading infectious cause of death after COVID-19. Apart from pulmonary involvement, which is the most common manifestation of TB, extrapulmonary TB (EPTB) affected 22.3% of TB patients in Hong Kong and was associated with a worse treatment outcome than pulmonary TB. Among EPTB, TB pleuritis (TBP) is the most prevalent form, accounting for 41.2% in Hong Kong and around 50% in two multi-centre Chinese studies.

Similar to other types of EPTB, the microbiological diagnosis of TBP is often difficult due to paucibacillary involvement (TB disease caused by a small number of bacteria) of the infected organs. Therefore, a significant proportion of patients received empirical anti-TB treatment based on compatible clinical presentations (exudative pleural effusion with raised adenosine deaminase level in pleural fluid), in the absence of diagnostic investigation results and alternative clinical explanation. The conventional diagnostic tests for TBP by acid-fast bacilli (AFB) stain and culture from the pleural fluid are insufficiently sensitive, and the long turnaround time of culture would delay the initial clinical management. Although a positive histological finding of granulomatous inflammation from the pleural biopsy is considered diagnostic equivalent for TBP, the procedural risk of pleural biopsy, especially bleeding and visceral injury is still a concern [9]. From the historical cohort of extrapulmonary TB in Hong Kong, only 10.6% and 39.7% of TBP were diagnosed by culture and histology respectively. Similarly, the efficacy of molecular tests on EPTB is also limited, presumably due to a low bacterial load and MTB DNA level. In a systematic review, the pooled sensitivity and specificity of Xpert® MTB/RIF (Xpert; Cepheid; Sunnyvale, CA, USA) on detecting MTB DNA in pleural fluid against culture were 50.9% and 99.2% in TBP. Given the low sensitivity, a negative Xpert result is not reliable to exclude TBP. The newest version of Xpert, Xpert® MTB/RIF Ultra (Xpert Ultra), was developed to improve the sensitivity of TB diagnosis and enhance rifampicin resistance identification. However, its diagnostic utility in TBP is still suboptimal. Mekkaoui et al reported the sensitivity and specificity of Xpert Ultra in the pleural fluid were 66.7% and 99.5% specificity. In another study comparing the diagnostic performance of Xpert Ultra and Xpert on EPTB by Christopher et al, Xpert Ultra had a higher sensitivity than Xpert (53.8% vs 46.2%) for pleural fluid against MTB culture and composite reference standard, but it did not reach statistical significance.

As a form of liquid biopsy, the MTB cell-free DNA (MTB cfDNA) in the pleural fluid may represent a rapid, novel and viable option to diagnose TBP. With this new tool, patients may not need to undergo a pleural biopsy to establish the diagnosis of TBP. Yang et al reported that the sensitivity of MTB cfDNA and Xpert was 79.5% and 38.5% respectively using the prespecified composite reference standard (incorporating the results of sputum culture, sputum Xpert, pleural effusion culture, pleural effusion Xpert or pleural biopsy), while the sensitivities would increase to 96.6% and 79.7% respectively in pleural fluid Xpert and/or culture-positive TBP samples. The reason for different sensitivities of MTB cfDNA in diagnosing TBP based on composite endpoints and microbiological methods was unclear, though it may be due to the different MTB bacterial load as reflected by the culture status in the pleural fluid. Nevertheless, this favourable result can be translated into the avoidance of more than 60% of unnecessary invasive pleural biopsies if MTB cfDNA is considered a gold standard for diagnosing TBP.

Before introducing the measurement of MTB cfDNA in diagnosing TBP, the correlation between MTB cfDNA level and MTB culture-positive TBP, MTB culture-negative TBP, and various types of non-TBP pleural effusion should be thoroughly evaluated. We hypothesize that the MTB cfDNA outperforms MTB culture in diagnosing TBP; with a high concordance rate between the MTB cfDNA level and the diagnosis of TBP, with high, intermediate and low MTB cfDNA levels in MTB culture-positive TBP, MTB culture-negative TBP, and non-TB pleural effusions respectively. Such concordance is a critical step to validate its diagnostic accuracy before introduction into the clinical setting.

The aim of the current study is to correlate the MTB cfDNA levels with various causes of pleural effusion and evaluate the diagnostic performance of different tests in diagnosing TBP.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized for unilateral pleural effusion.
* Pleural tapping will be performed for pleural fluid analysis.
* Aged 18 years old or above

Exclusion Criteria:

* History of tuberculous pleuritis (TBP) and bacterial pleural infection, in either ipsilateral or contralateral pleural space.
* History of intrapleural therapy (including talc and fibrinolytic) in the ipsilateral pleural space.
* History of surgical decortication or pleurodesis in the ipsilateral pleural space
* Use of anti-TB medications (including isoniazid, rifampicin, pyrazinamide, ethambutol, amikacin, streptomycin, levofloxacin, moxifloxacin, linezolid) for more than consecutive 14 days in the past 3 months.
* Failed to obtain informed consent due to patient's refusal or cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with definite or probably TBP will be recruited as positive control. Patients without TBP will be recruited as negative control.
Sampling Method: Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The MTB cfDNA level in TBP and non-TB pleural effusions | 24 months
  The median MTB cfDNA level in TBP and non-TB pleural effusions

SECONDARY OUTCOMES:
The diagnostic performance of MTB cfDNA and Xpert Ultra in diagnosing MTB culture-positive and MTB culture-negative TBP | 24 months
  Which includes sensitivity, specificity, positive predictive value, negative predictive value of these two tests in diagnosing TBP when comparing with the gold standard test
Clinical factors that may affect the levels of MTB cfDNA in TBP | 24 months
  which includes the mycobacterial culture result, level of inflammatory activity within the pleural space

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No